CLINICAL TRIAL: NCT04113421
Title: Quantitative 3-Dimensional Chest CT Vascular Reconstruction Before and After Anticoagulation for Pulmonary Embolism (OPTALYSE-3DAC)
Brief Title: Quantitative 3-Dimensional Chest CT Vascular Reconstruction Before and After Anticoagulation for Pulmonary Embolism
Acronym: OPTALYSE-3DAC
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Gregory Piazza, MD, MS, Associate Director, Thrombosis Research Group, Brigham and Women's Hospital
Other Study IDs: 2019P002124
Record Dates: First submitted 2019-10-01; First posted 2019-10-02 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Pulmonary Embolism
Keywords: pulmonary embolism; anticoagulation
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Anticoagulation: Inpatients diagnosed with acute PE, in whom clinical providers have elected to prescribe anticoagulation alone for treatment based on clinical grounds at BWH. In this population, a single follow-up contrast-enhanced chest CT will be performed to compare off-line with the contrast-enhanced chest CT done at baseline for the diagnosis of PE.
  Interventions: Diagnostic Test: Contrast-enhanced chest CT

INTERVENTIONS:
Diagnostic Test: Contrast-enhanced chest CT — A single follow-up contrast-enhanced chest CT to compare off-line with the contrast-enhanced chest CT done at baseline for the diagnosis of PE.

SUMMARY:
Design: U.S.-based, single-center, proof-of-concept study

Brief Description: A standard clinical contrast-enhanced chest CT scan performed 48 hours after clinically-indicated standard anticoagulation will be compared with a standard clinically-indicated baseline contrast-enhanced chest CT scan using a previously-studied and previously-validated 3-dimensional reconstruction technique to assess changes in the pulmonary vasculature in patients with acute pulmonary embolism (PE). This previously-studied and previously-validated 3-dimensional reconstruction technique has been used to assess the response of the pulmonary vasculature to catheter-based fibrinolysis in acute PE as well as to assess the pulmonary vasculature in a number of chronic lung diseases. However, the pulmonary vascular response to standard anticoagulation for acute PE has not been assessed previously.

Purpose: To compare the pulmonary vasculature before and after standard clinically-indicated anticoagulation for acute PE using a previously-studied and previously-validated 3-dimensional reconstruction technique applied with a standard clinically-indicated baseline contrast-enhanced chest CT scan (used to diagnose the acute PE) and a standard clinical contrast-enhanced chest CT scan performed 48 hours later as indicated by the study protocol.

Population: Inpatients diagnosed with acute PE, in whom clinical providers have prescribed standard anticoagulation alone for treatment based on clinical grounds at Brigham and Women's Hospital.

Enrollment: 10 subjects with acute PE

Clinical Site Location: Single-center, Brigham and Women's Hospital

Study Duration: 12 months

Primary Imaging Outcome: CT-determined percent change in perfusion of the pulmonary vasculature from baseline to 48 hours in inpatients diagnosed with acute PE, in whom clinical providers have prescribed standard anticoagulation alone for treatment based on clinical grounds at Brigham and Women's Hospital.

Secondary Imaging Outcome: CT-determined percent change in right ventricular (RV) volume from baseline to 48 hours in inpatients diagnosed with acute PE, in whom clinical providers have prescribed standard anticoagulation alone for treatment based on clinical grounds at Brigham and Women's Hospital.

DETAILED DESCRIPTION:
The pulmonary vascular response to ultrasound-facilitated, catheter-directed fibrinolysis for treatment of pulmonary embolism (PE) results in rapid improvement in patient symptoms and right ventricular (RV) recovery, while minimizing the risk of intracranial hemorrhage. The investigators recently completed an analysis of the chest computed tomographic (CT) data from the SEATTLE II Trial of ultrasound-facilitated, catheter-directed fibrinolysis for treatment of PE using a previously-validated 3-dimensional (3D) reconstruction technique pioneered at Brigham and Women's Hospital (BWH). This software-based 3D technique enables anatomic and structural resolution of the distal pulmonary arteries (microvasculature) far beyond the imaging capabilities of clinically utilized methods. This technique also provides a precise quantitation of RV volume and quantification of the perfusion of the proximal and distal pulmonary arteries. In our 3D reconstruction analysis of the multicenter, U.S.-based SEATTLE II Trial chest CT data, the investigators found that loss of intraparenchymal blood vessel volume was associated with RV enlargement and change in distal small vessel pulmonary artery perfusion predicted RV recovery with ultrasound-facilitated, catheter-directed fibrinolysis in subjects with acute PE. These data were presented at the American Heart Association (AHA) Annual Scientific Sessions in 2017 and have been submitted for publication.

While ultrasound-facilitated, catheter-directed fibrinolysis has been studied using this 3D reconstruction technique, the pulmonary vascular response in PE patients treated clinically with anticoagulation alone has not been. The investigators propose a study to evaluate inpatients diagnosed with acute PE, in whom clinical providers have already prescribed standard anticoagulation alone for treatment based on clinical grounds at Brigham and Women's Hospital, applying this 3-dimensional reconstruction technique to compare data from a standard clinical contrast-enhanced chest CT scan performed 48 hours after initiation of therapy and those data from the standard clinically-indicated baseline contrast-enhanced chest CT scan.

The specific aims for this proposed study are as follows:

Aim #1: To quantify the CT-determined percent change in perfusion of the pulmonary vasculature from baseline to 48 hours in inpatients diagnosed with acute PE, in whom clinical providers have prescribed standard anticoagulation alone for treatment based on clinical grounds at Brigham and Women's Hospital.

Hypothesis #1: The greatest change in pulmonary vascular perfusion following anticoagulation alone for acute PE will take place in the distal small (<5 mm2 cross-sectional area) pulmonary arteries compared with larger (>5 mm2 cross-sectional area) vessels. However, the magnitude of change will be less than that observed in our previously reported analysis focused on patients with acute PE undergoing ultrasound-facilitated, catheter-based fibrinolysis.

Aim #2: To quantify the CT-determined percent change in RV volume from baseline to 48 hours in inpatients diagnosed with acute PE, in whom clinical providers have prescribed standard anticoagulation alone for treatment based on clinical grounds at Brigham and Women's Hospital.

Hypothesis #2: RV volume will decrease over 48 hours of anticoagulation alone but the percent change will be less than that observed in our previously reported analysis focused on patients with acute PE undergoing ultrasound-facilitated, catheter-based fibrinolysis

ELIGIBILITY:
Inclusion Criteria:

* Inpatients diagnosed with acute PE, in whom clinical providers have elected to prescribe anticoagulation alone for treatment based on clinical grounds at BWH.
* Eligibility for the study will include patients over the age of 18 with bilateral proximal PE on CT (filling defect in ≥ 1 main, lobar, or segmental pulmonary artery), PE symptom duration ≤ 14 days, RV-to-LV diameter ratio ≥ 0.9 on contrast-enhanced chest CT, and a clinically-determined decision to pursue treatment with anticoagulation alone.

Exclusion Criteria:

1. Serum creatinine greater than 2 mg/dL
2. GFR < 60 mL/min
3. Pregnancy (pregnancy test will have been done as standardly required by Radiology before the initial clinically-indicated, clinically-protocolled chest CT)
4. Contrast allergy
5. Treatment with any fibrinolytics-based technique, or surgical/ catheter embolectomy
6. Expected hospital stay < 48 hours. The length of stay will be determined by the treating provider prior to enrollment. Subjects will not extend their stay to 48 hours if they are deemed ready for discharge prior to the time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients diagnosed with acute PE, in whom clinical providers have elected to prescribe anticoagulation alone for treatment based on clinical grounds at BWH.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Perfusion of the pulmonary arteries | 48 ± 6 hours
  Percent change in perfusion of the pulmonary arteries using quantitative 3-D vascular reconstruction of baseline and follow-up (at 48 ± 6 hours) standard contrast-enhanced chest CTs.

SECONDARY OUTCOMES:
Change in RV volume | 48 ± 6 hours
  Percent change in RV volume using quantitative 3-D vascular reconstruction of baseline and follow-up (at 48 ± 6 hours) standard contrast-enhanced chest CTs.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Piazza, MD, MS, Principal Investigator — BWH
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Will not participate in data sharing

REFERENCES:
- [Background] Tapson VF, Sterling K, Jones N, Elder M, Tripathy U, Brower J, Maholic RL, Ross CB, Natarajan K, Fong P, Greenspon L, Tamaddon H, Piracha AR, Engelhardt T, Katopodis J, Marques V, Sharp ASP, Piazza G, Goldhaber SZ. A Randomized Trial of the Optimum Duration of Acoustic Pulse Thrombolysis Procedure in Acute Intermediate-Risk Pulmonary Embolism: The OPTALYSE PE Trial. JACC Cardiovasc Interv. 2018 Jul 23;11(14):1401-1410. doi: 10.1016/j.jcin.2018.04.008. PMID 30025734
- [Background] Piazza G, Hohlfelder B, Jaff MR, Ouriel K, Engelhardt TC, Sterling KM, Jones NJ, Gurley JC, Bhatheja R, Kennedy RJ, Goswami N, Natarajan K, Rundback J, Sadiq IR, Liu SK, Bhalla N, Raja ML, Weinstock BS, Cynamon J, Elmasri FF, Garcia MJ, Kumar M, Ayerdi J, Soukas P, Kuo W, Liu PY, Goldhaber SZ; SEATTLE II Investigators. A Prospective, Single-Arm, Multicenter Trial of Ultrasound-Facilitated, Catheter-Directed, Low-Dose Fibrinolysis for Acute Massive and Submassive Pulmonary Embolism: The SEATTLE II Study. JACC Cardiovasc Interv. 2015 Aug 24;8(10):1382-1392. doi: 10.1016/j.jcin.2015.04.020. PMID 26315743